CLINICAL TRIAL: NCT01014104
Title: Administration of Methylprednisolone for Prevention of Ovarian Hyper Stimulation Syndrome in In-vitro Fertilization Cycles: A Randomized Controlled Trial
Brief Title: Administration of Methylprednisolone for Prevention of Ovarian Hyper Stimulation Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Hamid Gourabi, Chief, Royan Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Royan-Emb-005
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2009-11

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: Ovarian hyper stimulation syndrome; Methylprednisolone; IVF
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Case (Experimental): Administration of Methylprednisolone
  Interventions: Drug: Methylprednisolone
- Control (Sham Comparator)
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Methylprednisolone — Administration of Methylprednisolone
  Other Names: Case
  Arms: Case
Drug: Control — Normal salin injection
  Arms: Control

SUMMARY:
This study is a prospective randomized clinical controlled trial to assess the efficacy of the Methylprednisolone for preventing ovarian hyper stimulation syndrome in in vitro fertilization (IVF) cycles.

DETAILED DESCRIPTION:
Ovarian hyper stimulation syndrome is the most serious complication of ovarian stimulation which might be life threatening in the severe forms. Since there is still no definite cure for this syndrome, prevention is considered as an essential and vital issue. The objective of this study is to determine the effect of Methylprednisolone to prevent ovarian hyper stimulation syndrome in IVF cycles.

The study population comprises all infertile patients with diagnosis of polycystic ovarian syndrome which will undergo of in-vitro fertilization. The PCO subjects will be recognized based on the Rotterdam criteria inclusive the presence of least 2 signs of oligomenorrhea, hyper androgynism (clinical or laboratory), LH/FSH>2 and ovarian morphological evidences in Doppler ultrasound.

The existence of more than 20 follicles in both ovaries and E2 concentration >4000 pg/ml will be considered as the OHSS risk factors.

In this study all eligible patients will be randomly allocated into two study groups by a computerized randomization method:

Treatment group (case) will be administered 16 mg Methylprednisolone initiated from the first day of stimulation and will be tapered after the first pregnancy test (day 13 after the embryo transfer). Furthermore, these patients will receive a bolus IV dose methylprednisolone, 1g on the day of egg collection and embryo transfer.

Patients in the control group will not receive any treatment with glucocorticoids. If each group confronts with every kind of high risk signs or symptoms, they will undergo coasting or gonadotropin withdrawal or other treatment strategies.

The presence of OHSS is defined in accordance with the Golan 5 grade system and women who at least are at grade 2 of this classification (Mild) considered as OHSS cases and will experience abdominal distention and discomfort, nausea and vomiting and/or diarrhea and enlargement of ovaries(5-12cm). In Moderate forms, ultrasound evidences of ascites will be observed and severe OHSS accompany with clinical signs of ascites, hydrothorax, breathing disorders, hemoconcentration, coagulopathy and renal perfusion decrease.

ELIGIBILITY:
Inclusion Criteria:

* Poly Cystic Ovarian Syndrome patients
* Indication for IVF/ICSI and Long Protocol ovarian stimulation
* Basal FSH≥10
* Normal BMI (20-25)
* physical health

Exclusion Criteria:

* Allergy to GnRH analogues, FSH and corticosteroids
* presence of heart failure, recent myocardial infarction
* Hypertension
* Diabetes mellitus
* epilepsy
* glaucoma
* hypothyroidism
* hepatic failure
* osteoporosis
* peptic ulceration
* renal impairment
* Using drugs that have interaction with corticosteroids such

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2009-10; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Occurrence rate of Ovarian hyper stimulation syndrome | Until 20 days after embryos transfer

SECONDARY OUTCOMES:
Estradiol concentration in the day before hCG administration | Until 20 days after embryos transfer
Retrieved and injected oocytes number and quality | Until 20 days after embryos transfer
Achieved and transferred embryos number and quality | Until 20 days after embryos transfer
Implantation rate | Until 20 days after embryos transfer
Chemical and clinical pregnancy rate and cancelation rate | Until 20 days after embryos transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Moini, MD, Principal Investigator — Endocrinology and Female Infertility Department, Reproductive Medicine Research Center, Royan institute, ACECR, Tehran, Iran; Marzieh Shiva, MD, Principal Investigator — Endocrinology and Female Infertility Department, Reproductive Medicine Research Center, Royan institute, ACECR, Tehran, Iran; Narges bagheri lankarani, MD, Principal Investigator — Endocrinology and Female Infertility Department, Reproductive Medicine Research Center, Royan institute, ACECR, Tehran, Iran
Locations (1):
- Royan Institute, Tehran, Tehran Province, Iran

REFERENCES:
- See also: Related Info — http://www.royaninstitute.org